CLINICAL TRIAL: NCT04631822
Title: Comparative Study Between Dexamethasone, and Dexmedetomidine as Additives to Bupivacaine in Ultrasound Guided Adductor Canal Block in Knee Arthroscopy
Brief Title: Comparing Dexamethasone With Dexmedetomidine as Additives to Bupivacaine in Adductor Canal Block for Knee Arthroscopy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rasha Hamed (Other)
Responsible Party: Sponsor-Investigator, Rasha Hamed, Rasha Hamed, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: knee regional anaesthesia
Record Dates: First submitted 2020-10-26; First posted 2020-11-17 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Pain, Postoperative
Keywords: adductor canal regional block; anaesthesia for knee arthroscopic surgeries
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Spinal; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexamethasone, combined with bupivacaine for adductor canal block (Active Comparator): All patients will receive spinal anesthesia with 3 ml 0.5% hyperbaric bupivacaine at the L3/4 interspaces in the setting position. Ultrasound blocks will be done immediately after spinal anesthesia, before surgical intervention.
  In this arm, patients will receive 20 ml mixture of 0.25% bupivacaine and 8 mg dexamethasone.
  Interventions: Procedure: Spinal anaesthesia; Procedure: ultrasound-guided Adductor Canal Block + dexamethasone
- Dexmedetomedine, combined with bupivacaine for adductor canal block (Active Comparator): All patients will receive spinal anesthesia with 3 ml 0.5% hyperbaric bupivacaine at the L3/4 interspaces in the setting position. Ultrasound blocks will be done immediately after spinal anesthesia, before surgical intervention.
  In this arm, patients will receive 20 ml mixture of 0.25% bupivacaine and 0.5 Mg/kg dexmedetomidine.
  Interventions: Procedure: Spinal anaesthesia; Procedure: ultrasound-guided Adductor Canal Block + dexmedetomedine
- control group (Active Comparator): All patients will receive spinal anesthesia with 3 ml 0.5% hyperbaric bupivacaine at the L3/4 interspaces in the setting position. Ultrasound blocks will be done immediately after spinal anesthesia, before surgical intervention.
  In this arm, patients will receive 20 ml mixture of 0.25% bupivacaine with no additives
  Interventions: Procedure: ultrasound-guided Adductor Canal Block

INTERVENTIONS:
Procedure: Spinal anaesthesia — spinal anesthesia shall be conducted with 2.5 ml 0.5% hyperbaric bupivacaine at the L3/4 interspaces in the setting position.
  Arms: Dexamethasone, combined with bupivacaine for adductor canal block; Dexmedetomedine, combined with bupivacaine for adductor canal block
Procedure: ultrasound-guided Adductor Canal Block + dexamethasone — Ultrasound blocks will be done immediately after spinal anesthesia, before surgical intervention. A high-frequency linear ultrasound transducer was placed transverse to the longitudinal axis of the extremity at the midthigh level at a distance approximately halfway between the iliac spine and the patella. The femoral artery was identified underneath the sartorius muscle with the vein just underneath the artery. At this position, the saphenous nerve was placed lateral to the artery in the adductor canal (Fig. 1). A 10 cm Tuohy canula 18G "Gauge" (Braun Medical, Melsungen, Germany) was inserted, in plane, from the lateral side of the transducer, through the sartorius muscle with the tip placed lateral to the artery. then, a 20-ml mixture of 0.25% bupivacaine, and 4 mg dexamethasone will be injected.
  Arms: Dexamethasone, combined with bupivacaine for adductor canal block
Procedure: ultrasound-guided Adductor Canal Block + dexmedetomedine — Ultrasound blocks will be done immediately after spinal anesthesia, before surgical intervention. A high-frequency linear ultrasound transducer was placed transverse to the longitudinal axis of the extremity at the midthigh level at a distance approximately halfway between the iliac spine and the patella. The femoral artery was identified underneath the sartorius muscle with the vein just underneath the artery. At this position, the saphenous nerve was placed lateral to the artery in the adductor canal (Fig. 1). A 10 cm Tuohy canula 18G "Gauge" (Braun Medical, Melsungen, Germany) was inserted, in plane, from the lateral side of the transducer, through the sartorius muscle with the tip placed lateral to the artery.then, a 20-ml mixture of 0.25% bupivacaine, and 0.5 Mg/kg dexmedetomidine will be injected.
  Arms: Dexmedetomedine, combined with bupivacaine for adductor canal block
Procedure: ultrasound-guided Adductor Canal Block — Ultrasound blocks will be done immediately after spinal anesthesia, before surgical intervention. A high-frequency linear ultrasound transducer was placed transverse to the longitudinal axis of the extremity at the midthigh level at a distance approximately halfway between the iliac spine and the patella. The femoral artery was identified underneath the sartorius muscle with the vein just underneath the artery. At this position, the saphenous nerve was placed lateral to the artery in the adductor canal (Fig. 1). A 10 cm Tuohy canula 18G "Gauge" (Braun Medical, Melsungen, Germany) was inserted, in plane, from the lateral side of the transducer, through the sartorius muscle with the tip placed lateral to the artery.then, a 20-ml mixture of 0.25% bupivacaine
  Arms: control group

SUMMARY:
a comparison shall be conducted between dexamethasone accompanied by bupivacaine, on one hand, and dexmedetomedine accompanied by bupivacaine on the other hand and a control group for pain-free knee arthroscopic surgeries.

DETAILED DESCRIPTION:
Arthroscopic knee surgery can cause significant postoperative pain to the degree that can potentially delay timely discharge from the ambulatory surgical setting. Analgesia after knee surgery can be provided by multiple, non-systemic, non-opioid-based methods, including local anesthetic infiltration, peripheral nerve blockade, neuraxial procedures, and intra-articular injections. The femoral nerve block has been shown to be superior to traditional intra-articular injection of local anesthetics in some knee surgeries, but motor blockade of the quadriceps muscle, with the potential risk for falls, limits the value of femoral blocks for less invasive ambulatory surgery. Orthopedic surgery is increasingly being performed on an ambulatory basis, where perioperative analgesia can improve timely discharge in the outpatient setting.

ELIGIBILITY:
Inclusion Criteria: -

* Adult patients of aged more than 18 years old ASA "American Society of Anaesthesia"
* physical status I or II under-going any unilateral knee arthroscopy. Exclusion Criteria: -
* patient refusal.
* Pre-existing pain ; postoperative pain similar to preoperative pain
* Known contraindications to peripheral nerve block, including local skin infections, bleeding diathesis, and coagulopathy.
* Allergies to local anesthetics, dexmedetomidine, or any component of multimodal analgesia.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Dynamic Visual Analogue Scale score | month 1 postoperative
  a scale of 11 points. 0 = no pain, 10=worst pain

SECONDARY OUTCOMES:
Dynamic Visual Analogue Scale score | month 3 postoperative
  a scale of 11 points. 0 = no pain, 10=worst pain
24 hours opioid analgesia consumed | 24 hours postoperative
Visual Analogue Scale score | 24 hours postoperative
  a scale of 11 points. 0 = no pain, 10=worst pain
month 3 opioid analgesia | month 3 postoperative
  amount of oral codeine consumed postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy A Yousef, MD, Study Chair — Professor of Anesthesia and Intensive care unit, faculty of medicine, Assiut University; yara A yousef, Lecturer, Study Director — Lecturer of Anesthesia and Intensive care unit, faculty of medicine, Assiut University; rasha hamed, MD, Principal Investigator — aisstant professor of anesthesia and ICU
Locations (1):
- Rasha Hamed, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iskandar H, Benard A, Ruel-Raymond J, Cochard G, Manaud B. Femoral block provides superior analgesia compared with intra-articular ropivacaine after anterior cruciate ligament reconstruction. Reg Anesth Pain Med. 2003 Jan-Feb;28(1):29-32. doi: 10.1053/rapm.2003.50019. PMID 12567340
- [Background] Ilfeld BM, Duke KB, Donohue MC. The association between lower extremity continuous peripheral nerve blocks and patient falls after knee and hip arthroplasty. Anesth Analg. 2010 Dec;111(6):1552-4. doi: 10.1213/ANE.0b013e3181fb9507. Epub 2010 Oct 1. PMID 20889937
- [Background] Fortier J, Chung F, Su J. Unanticipated admission after ambulatory surgery--a prospective study. Can J Anaesth. 1998 Jul;45(7):612-9. doi: 10.1007/BF03012088. PMID 9717590
- [Background] Akkaya T, Ersan O, Ozkan D, Sahiner Y, Akin M, Gumus H, Ates Y. Saphenous nerve block is an effective regional technique for post-menisectomy pain. Knee Surg Sports Traumatol Arthrosc. 2008 Sep;16(9):855-8. doi: 10.1007/s00167-008-0572-4. Epub 2008 Jun 24. PMID 18574578
- [Background] Kapoor R, Adhikary SD, Siefring C, McQuillan PM. The saphenous nerve and its relationship to the nerve to the vastus medialis in and around the adductor canal: an anatomical study. Acta Anaesthesiol Scand. 2012 Mar;56(3):365-7. doi: 10.1111/j.1399-6576.2011.02645.x. PMID 22335278
- [Background] Horn JL, Pitsch T, Salinas F, Benninger B. Anatomic basis to the ultrasound-guided approach for saphenous nerve blockade. Reg Anesth Pain Med. 2009 Sep-Oct;34(5):486-9. doi: 10.1097/AAP.0b013e3181ae11af. PMID 19920424
- [Background] Benzon HT, Sharma S, Calimaran A. Comparison of the different approaches to saphenous nerve block. Anesthesiology. 2005 Mar;102(3):633-8. doi: 10.1097/00000542-200503000-00023. PMID 15731603
- [Background] Manickam B, Perlas A, Duggan E, Brull R, Chan VW, Ramlogan R. Feasibility and efficacy of ultrasound-guided block of the saphenous nerve in the adductor canal. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):578-80. doi: 10.1097/aap.0b013e3181bfbf84. PMID 19916251
- [Background] Ishiguro S, Yokochi A, Yoshioka K, Asano N, Deguchi A, Iwasaki Y, Sudo A, Maruyama K. Technical communication: anatomy and clinical implications of ultrasound-guided selective femoral nerve block. Anesth Analg. 2012 Dec;115(6):1467-70. doi: 10.1213/ANE.0b013e31826af956. Epub 2012 Aug 10. PMID 22886842
- [Background] Lund J, Jenstrup MT, Jaeger P, Sorensen AM, Dahl JB. Continuous adductor-canal-blockade for adjuvant post-operative analgesia after major knee surgery: preliminary results. Acta Anaesthesiol Scand. 2011 Jan;55(1):14-9. doi: 10.1111/j.1399-6576.2010.02333.x. Epub 2010 Oct 29. PMID 21039357
- [Background] Horner G, Dellon AL. Innervation of the human knee joint and implications for surgery. Clin Orthop Relat Res. 1994 Apr;(301):221-6. PMID 8156678
- [Background] Jenstrup MT, Jaeger P, Lund J, Fomsgaard JS, Bache S, Mathiesen O, Larsen TK, Dahl JB. Effects of adductor-canal-blockade on pain and ambulation after total knee arthroplasty: a randomized study. Acta Anaesthesiol Scand. 2012 Mar;56(3):357-64. doi: 10.1111/j.1399-6576.2011.02621.x. Epub 2012 Jan 4. PMID 22221014
- [Background] An K, Elkassabany NM, Liu J. Dexamethasone as adjuvant to bupivacaine prolongs the duration of thermal antinociception and prevents bupivacaine-induced rebound hyperalgesia via regional mechanism in a mouse sciatic nerve block model. PLoS One. 2015 Apr 9;10(4):e0123459. doi: 10.1371/journal.pone.0123459. eCollection 2015. PMID 25856078
- [Background] Abdallah FW, Dwyer T, Chan VW, Niazi AU, Ogilvie-Harris DJ, Oldfield S, Patel R, Oh J, Brull R. IV and Perineural Dexmedetomidine Similarly Prolong the Duration of Analgesia after Interscalene Brachial Plexus Block: A Randomized, Three-arm, Triple-masked, Placebo-controlled Trial. Anesthesiology. 2016 Mar;124(3):683-95. doi: 10.1097/ALN.0000000000000983. PMID 26649424
- [Background] Kaur M, Singh PM. Current role of dexmedetomidine in clinical anesthesia and intensive care. Anesth Essays Res. 2011 Jul-Dec;5(2):128-33. doi: 10.4103/0259-1162.94750. PMID 25885374
- [Derived] Elsawy S, Abdelwahab A, Hamdi Y, Hamed RAA. Dexamethasone as an additive to bupivacaine in an ultrasound-guided adductor canal block for the management of persistent pain after arthroscopic reconstruction of the anterior cruciate ligament: a randomized, double-blind study. BMC Anesthesiol. 2025 Apr 24;25(1):208. doi: 10.1186/s12871-025-02921-6. PMID 40275160